CLINICAL TRIAL: NCT05748717
Title: The Relationship of Transcranial Doppler Velocity With Other Vascular Measurements in Children With Sickle Cell Anaemia
Brief Title: Arterial Function Parameters and Transcranial Doppler Velocity in Paediatric Patients With Sickle Cell Disease
Acronym: AFAT
Status: Recruiting | Type: Observational
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Marvin E Reid, Professor, The University of The West Indies
Other Study IDs: CREC-MN.88/2020/2021
Record Dates: First submitted 2023-02-05; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell disease; Transcranial Doppler Velocity; Arterial Stiffness; Augmentation Index; Arterial Function
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paediatric patients with sickle cell disease with normal TCD velocity without clinical stroke: Patients in this group will be aged 4 to 16 years with sickle cell anaemia with no prior history of stroke or previous Transcranial Doppler study showing a maximum time-averaged mean velocity of greater than 169 cm/sec, and who have not received a red cell transfusion in the past two months and are considered to be at steady state.
- Paediatric patients with sickle cell disease with an abnormal TCD velocity (with or without stroke): Patients in this group will be aged 4 to 16 years with sickle cell anaemia with an abnormal TCD velocity, who have not received a red cell transfusion in the past two months and are considered to be at steady state.

SUMMARY:
Structural and functional changes in arteries are increasingly being recognized as significant features of sickle cell disease. This study aims to determine whether there are differences in arterial function parameters between children with sickle cell disease with normal and abnormal transcranial Doppler velocity. After informed consent is obtained, participants will have vascular, Transcranial Doppler, haematological and biochemical parameters measured. Researchers will compare children with sickle cell disease who have normal Transcranial Doppler velocity and no history of stroke with children with those who have an abnormal Transcranial Doppler velocity with or without a history of stroke to see if there are significant differences in arterial function parameters.

DETAILED DESCRIPTION:
Structural and functional changes in arteries are increasingly being recognized as significant features of sickle cell disease and arterial function in sickle cell anaemia (SCA) is gaining importance.

The goal of this observational study is to compare arterial parameters in children with sickle cell disease who have normal or abnormal Transcranial Doppler velocity. The main question it aims to answer is: whether there is a significant difference in arterial Function parameters measured by aortic pulse wave velocity, augmentation index, brachial and central blood pressure in Jamaican children with Sickle Cell anaemia who attend the Sickle Cell Unit in Kingston Jamaica who are reported to have normal or an abnormal Transcranial Doppler velocity and whether the probability of having an abnormal Transcranial Doppler velocity or higher arterial function parameters is increased by specific biophysical markers.

Participants who are identified will be informed about the study and potential risks. All patients giving written informed consent will then undergo arterial function (arteriograph,TensioMed® Arteriograph24™,Budapest, H-1181 Hungary), Transcranial Doppler, haematological and biochemical measurements.

Researchers will compare children with sickle cell disease who have normal Transcranial Doppler velocity and no history of stroke with children with this illness who have an abnormal Transcranial Doppler velocity to see if there are significant differences in regional arterial function.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric participants with sickle cell anaemia (HbSS, HbSβ0 thalassemia, HbSD, HbSOArab)
2. Age: Between 4-16 years of age, at the time of enrolment
3. Has had at least one complete TCD study whether or not on hydroxyurea treatment or in a clinical trial.
4. Parent or guardian willing and able to provide informed consent and child gives assent
5. Ability to comply with study-related evaluations.

Exclusion Criteria:

* Participants who meet any of the following criteria are disqualified from enrollment in the study:

  1. Patients in whom a TCD study cannot be completed
  2. Patients who have had an Erythrocyte transfusion in the past two months
  3. Patients who are acutely ill or have had an acute infection in the past two weeks

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric participants with sickle cell anemia (HbSS, HbSβ0 thalassemia, HbSD, HbSOArab) Age 4-16 years with or without a previous stroke with at least one previous transcranial Doppler study.
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean difference in aortic pulse wave velocity in mmHg between patients with an abnormal transcranial Doppler Velocity compared to those with a normal Transcranial Doppler velocity without stroke | Three measurements will be taken over 10 minutes at the study visit.
  The primary outcome of aortic pulse wave velocity in mmHg, will be measured in all patients with an Arteriograph 24 (TensioMed, Budapest, Hungary). Before the assessment, the patient will be allowed to rest for 5 -10 minutes. An appropriate cuff size will be used for each patient. The test will be carried out in a calm, temperature-controlled room.
Mean difference in aortic augmentation index, in % between patients with an abnormal transcranial Doppler Velocity compared to those with a normal Transcranial Doppler velocity without stroke. | Three measurements will be taken over 10 minutes at the study visit.
  The primary outcome of aortic augmentation index, in % will be measured in all patients with an Arteriograph 24 (TensioMed, Budapest, Hungary). Before the assessment, the patient will be allowed to rest for 5 -10 minutes. An appropriate cuff size will be used for each patient. The test will be carried out in a calm, temperature-controlled room.

SECONDARY OUTCOMES:
Mean difference in brachial augmentation index, in %, between patients with an abnormal transcranial Doppler Velocity compared to those with a normal Transcranial Doppler velocity without stroke | Three measurements will be taken over 10 minutes at the study visit.
  Brachial augmentation index, in %, will be measured in all patients with an Arteriograph 24 (TensioMed, Budapest, Hungary). Before the assessment, the patient will be allowed to rest for 5 -10 minutes. An appropriate cuff size will be used for each patient. The test will be carried out in a calm, temperature-controlled room.
Mean difference in aortic systolic blood pressure in mmHg between patients with an abnormal transcranial Doppler Velocity compared to those with a normal Transcranial Doppler velocity without stroke | Three measurements will be taken over 10 minutes at the study visit.
  Aortic systolic blood pressure in mmHg, will be measured in all patients with an Arteriograph 24 (TensioMed, Budapest, Hungary). Before the assessment, the patient will be allowed to rest for 5 -10 minutes. An appropriate cuff size will be used for each patient. The test will be carried out in a calm, temperature-controlled room.
Mean difference in aortic pulse pressure, in mmHg between patients with an abnormal transcranial Doppler Velocity compared to those with a normal Transcranial Doppler velocity without stroke | Three measurements will be taken over 10 minutes at the study visit.
  Aortic pulse pressure in mmHg, will be measured in all patients with an Arteriograph 24 (TensioMed, Budapest, Hungary). Before the assessment, the patient will be allowed to rest for 5 -10 minutes. An appropriate cuff size will be used for each patient. The test will be carried out in a calm, temperature-controlled room.
Mean difference in brachial systolic pressure in mmHg, between patients with an abnormal transcranial Doppler Velocity compared to those with a normal Transcranial Doppler velocity without stroke | Three measurements will be taken over 10 minutes at the study visit.
  Brachial systolic pressure in mmHg will be measured in all patients with an Arteriograph 24 (TensioMed, Budapest, Hungary). Before the assessment, the patient will be allowed to rest for 5 -10 minutes. An appropriate cuff size will be used for each patient. The test will be carried out in a calm, temperature-controlled room.
Mean difference in brachial diastolic pressure in mmHg between patients with an abnormal transcranial Doppler Velocity compared to those with a normal Transcranial Doppler velocity without stroke. | Three measurements will be taken over 10 minutes
  Brachial diastolic pressure in mmHg will be measured in all patients with an Arteriograph 24 (TensioMed, Budapest, Hungary). Before the assessment, the patient will be allowed to rest for 5 -10 minutes. An appropriate cuff size will be used for each patient. The test will be carried out in a calm, temperature-controlled room.
Difference in mean arterial pressure in mmHg between patients with an abnormal transcranial Doppler Velocity compared to those with a normal Transcranial Doppler velocity without stroke | Three measurements will be taken over 10 minutes
  Mean arterial pressure in mmHg will be measured in all patients with an Arteriograph 24 (TensioMed, Budapest, Hungary). Before the assessment, the patient will be allowed to rest for 5 -10 minutes. An appropriate cuff size will be used for each patient. The test will be carried out in a calm, temperature-controlled room.

CONTACTS AND LOCATIONS:
Locations (1):
- Caribbean Institute for Health Research, The University of the West Indies, Kingston, Saint Andrew Parish, Jamaica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palomarez A, Jha M, Medina Romero X, Horton RE. Cardiovascular consequences of sickle cell disease. Biophys Rev (Melville). 2022 Aug 8;3(3):031302. doi: 10.1063/5.0094650. eCollection 2022 Sep. PMID 38505276
- [Background] Ranque B, Menet A, Boutouyrie P, Diop IB, Kingue S, Diarra M, N'Guetta R, Diallo D, Diop S, Diagne I, Sanogo I, Tolo A, Chelo D, Wamba G, Gonzalez JP, Abough'elie C, Diakite CO, Traore Y, Legueun G, Deme-Ly I, Faye BF, Seck M, Kouakou B, Kamara I, Le Jeune S, Jouven X. Arterial Stiffness Impairment in Sickle Cell Disease Associated With Chronic Vascular Complications: The Multinational African CADRE Study. Circulation. 2016 Sep 27;134(13):923-33. doi: 10.1161/CIRCULATIONAHA.115.021015. Epub 2016 Aug 31. PMID 27582423
- [Background] Hulbert ML, McKinstry RC, Lacey JL, Moran CJ, Panepinto JA, Thompson AA, Sarnaik SA, Woods GM, Casella JF, Inusa B, Howard J, Kirkham FJ, Anie KA, Mullin JE, Ichord R, Noetzel M, Yan Y, Rodeghier M, Debaun MR. Silent cerebral infarcts occur despite regular blood transfusion therapy after first strokes in children with sickle cell disease. Blood. 2011 Jan 20;117(3):772-9. doi: 10.1182/blood-2010-01-261123. Epub 2010 Oct 12. PMID 20940417
- [Background] Belizna C, Loufrani L, Ghali A, Lahary A, Primard E, Louvel JP, Henrion D, Levesque H, Ifrah N. Arterial stiffness and stroke in sickle cell disease. Stroke. 2012 Apr;43(4):1129-30. doi: 10.1161/STROKEAHA.111.635383. Epub 2011 Dec 22. PMID 22198986
- [Background] Lemogoum D, Van Bortel L, Najem B, Dzudie A, Teutcha C, Madu E, Leeman M, Degaute JP, van de Borne P. Arterial stiffness and wave reflections in patients with sickle cell disease. Hypertension. 2004 Dec;44(6):924-9. doi: 10.1161/01.HYP.0000148506.73622.ba. Epub 2004 Nov 8. PMID 15534075
- [Background] Pikilidou M, Yavropoulou M, Antoniou M, Papakonstantinou E, Pantelidou D, Chalkia P, Nilsson P, Yovos J, Zebekakis P. Arterial Stiffness and Peripheral and Central Blood Pressure in Patients With Sickle Cell Disease. J Clin Hypertens (Greenwich). 2015 Sep;17(9):726-31. doi: 10.1111/jch.12572. Epub 2015 May 20. PMID 25991400
- [Background] Adams RJ, Nichols FT, Figueroa R, McKie V, Lott T. Transcranial Doppler correlation with cerebral angiography in sickle cell disease. Stroke. 1992 Aug;23(8):1073-7. doi: 10.1161/01.str.23.8.1073. PMID 1636180